CLINICAL TRIAL: NCT03316963
Title: Local Neostigmine for Treatment of Snoring During Drug-Induced Sleep Endoscopy
Brief Title: Neostigmine For Snoring During DISE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI is moving the a new institution and ended the study early.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Raj Dedhia, Asstant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00096770
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Snoring
Keywords: Neostigmine; Nerve stimulant medication; Treatments for snoring
MeSH Terms: conditions — Snoring | interventions — Neostigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug-induced sleep endoscopy (DISE) with Neostigmine (Experimental): Artificial sleep will be induced by intravenous administration of propofol with micro boluses until clinical sleep is achieved with spontaneous respiration and observed apneas under monitored anesthesia care. Endoscopy will be performed with visualization on a monitor and recording on a digital recorder. After the patient demonstrates snoring and obstruction collapse, the patient will receive the study medication (neostigmine methylsulfate 1mg/mL) into the soft palate.
  Interventions: Drug: Neostigmine Methylsulfate

INTERVENTIONS:
Drug: Neostigmine Methylsulfate — After the patient demonstrates snoring and obstruction collapse, the patient will receive the study medication (neostigmine methylsulfate 1mg/mL) into the soft palate with co-administration of intravenous glycopyrrolate 0.2mg. At each of 5 injection sites on the soft palate , 0.5 mL (0.5mg) of neostigmine methylsulfate will be administered, yielding a total of 2.5mg (2.5mL) of neostigmine methylsulfate. The medication will be administered using five 1 mL syringes filled with 0.5 mL neostigmine each. Following administration of neostigmine, the patient will be observed for an additional 4 minutes to examine both vibration and sound emanating from the soft palate. The anticipated time under sedation will be 14 minutes.

SUMMARY:
The study team is seeking a novel treatment for snoring involving local application of a nerve stimulant medication, neostigmine. In this study, neostigmine will be injected into 5 sites of the soft palate during a standard procedure, drug-induced sleep endoscopy, to evaluate the effect on snoring.

DETAILED DESCRIPTION:
Snoring is a major problem, affecting 40 million Americans. The disease affects patient and partner sleep quality as well as daytime function. Snoring treatment is limited by device compliance (mouth appliance, positive airway pressure) and insurance does not regularly pay for these devices. Surgical treatment for snoring has mixed results. As a result, there is an important need to develop new treatments for snoring.

The study team is seeking a novel treatment for snoring involving local application of a nerve stimulant medication, neostigmine. In this study, neostigmine will be injected into 5 sites of the soft palate during a standard procedure, drug-induced sleep endoscopy, to evaluate the effect on snoring. If successful, development of a topical (non-injectable) version of this drug will be considered, so that the patient can apply him/herself before bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Snoring or mild obstructive sleep apnea
* English-speaking
* Greater than 18 years old
* Able to give informed consent

Exclusion Criteria:

* On active anti-coagulation medication
* Pregnant women
* Hypersensitivity to neostigmine
* Peritonitis or mechanical obstruction of the intestinal or urinary tract
* Coronary artery disease
* Cardiac arrhythmia
* Recent acute coronary syndrome
* Myasthenia gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Change in decibel sound after injection of neostigmine | The DISE will occur up to 30 days after the pre-op visit and study enrollment
  The data will come from the drug-induced sleep endoscopy (DISE) audio and video recordings. Prior to the neostigmine injection, a snoring microphone will be placed over the right clavicle. Following administration of neostigmine, the patient will be observed for an additional 4 minutes to examine sound emanating from the soft palate. Total run time, instantaneous decibel levels, LAeq (average decibel level over time), and the maximum decibel level will be recorded.
Change in soft palate motion after injection of neostigmine | The DISE will occur up to 30 days after the pre-op visit and study enrollment
  The data will come from the drug-induced sleep endoscopy (DISE) audio and video recordings. Following administration of neostigmine, the patient will be observed for an additional 4 minutes to examine vibration emanating from the soft palate.

CONTACTS AND LOCATIONS:
Overall Officials: Raj C. Dedhia, MD MS, Principal Investigator — Emory University
Locations (1):
- Raj C. Dedhia, Atlanta, Georgia, United States